CLINICAL TRIAL: NCT05455866
Title: Central Venous Catheter-related Complications in Patients Under Anticancer Treatment: a Prospective Monocentric Study on Incidence and Consequences
Brief Title: Central Venous Catheter-related Complications in Patients Under Anticancer Treatment
Acronym: KTcCHO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Alpes Leman (Other)
Responsible Party: Sponsor
Other Study IDs: KTcCHO
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Central Venous Catheter Thrombosis; Central Venous Catheter Related Bloodstream Infection; Solid Tumor; Hematologic Malignancy
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis; Hematologic Neoplasms | interventions — Central Venous Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: central venous catheter — collection and descriptionof central venous catheter-related complications

SUMMARY:
Oncology and hemotology patients under anticancer treatments are exposed to increased risks of central venous catheter-related complications due to the underlying cancer and its treament.

This prospective observational monocentric french study aims at describing the incidence of such complications, their morbimortality, and analyzing some risk factors in order to contribute to propose some strategies to reduce these complications' rate and consequences

ELIGIBILITY:
Inclusion Criteria:

All patients older than 18 years, with solid cancer or hematological malignancy receiving anticancer treatment in the outpatient medical department of Alpes Leman Hospital and having a central venous catheter been placed between the 11th of July 2022, and the 1st of January 2023.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients at Oncohematology Outpatient Department
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-11 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate and density of central venous catheter-related complications (infections, thromboses, extravasation) | 6 months

SECONDARY OUTCOMES:
Incidence rate of severe central venous catheter-related complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence OBERKAMPF, Principal Investigator — Centre Hospitalier Alpes Leman